CLINICAL TRIAL: NCT02744625
Title: Physiologic Study of Cerebral Perfusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Responsible Party: Principal Investigator, François Lamontagne, Clinician Scientist, Université de Sherbrooke
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2016-1267
Record Dates: First submitted 2016-04-07; First posted 2016-04-20 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Cerebral Perfusion Pressure; Vasopressor Agents; Shock; Magnetic Resonance Imaging (MRI), Functional
MeSH Terms: conditions — Shock | interventions — Propofol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Shock lower Mean Arterial Pressure (MAP) (Active Comparator): Vasopressor-dependent treated to lower MAP (65 mmHg)
  Interventions: Drug: Lower doses of vasopressor therapy for a MAP of 65 mmHg; Drug: Propofol for light sedation
- Shock higher MAP (Experimental): Vasopressor-dependent treated to higher MAP (75 mmHg)
  Interventions: Drug: Higher doses of vasopressor therapy for a MAP of 75 mmHg; Drug: Propofol for light sedation
- Healthy participant awake (No Intervention): Healthy participant awake
- Healthy participant sedated (Experimental): Healthy participant Under light sedation
  Interventions: Drug: Propofol for light sedation

INTERVENTIONS:
Drug: Higher doses of vasopressor therapy for a MAP of 75 mmHg
  Arms: Shock higher MAP
Drug: Lower doses of vasopressor therapy for a MAP of 65 mmHg
  Arms: Shock lower Mean Arterial Pressure (MAP)
Drug: Propofol for light sedation — Propofol for light sedation
  Arms: Healthy participant sedated; Shock higher MAP; Shock lower Mean Arterial Pressure (MAP)

SUMMARY:
The aim of the study is to measure cerebral perfusion using MRI in healthy subjects (with and without sedation) and in vasopressor-dependent patients

ELIGIBILITY:
Healthy Subjects :

* Inclusion criteria :

  * being over 18 years old
* Exclusion criterias :

  * having a positive serum pregnancy test
  * having a contraindication to MRI
  * having a contraindication to receive light sedation with propofol
  * suffering of claustrophobia or of anxiety disorder

Shock Subjects :

* Inclusion criterias :

  * being over 18 years old
  * being hospitalized to the medical intensive care unit of the CHUS Fleurimont
  * being in a stabilized shock state, primarily of distributive etiology
  * having received an appropriate fluid resuscitation, as judged by the attending physician
* Exclusion criterias :

  * having a different primary etiology of shock than distributive (cardiogenic, hypovolemic, obstructive)
  * needing vasopressor therapy as the result of extracorporeal circulation
  * having known cerebral lesions
  * having an intra-aortic balloon pump
  * being in a palliative or near end-of-life situation
  * having a contraindication to MRI
  * suffering of claustrophobia or of anxiety disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-04; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Global and regional cerebral blood flow | Within 15 minutes of intervention initiation
  Cerebral blood flow will be measured by the arterial spin labeling technique (ASL) which provides information expressed in mL/100g/min. Using 3-T MRI technology,we will first acquire T1 images of the brain and sub-regions of interest. Thereafter, ASL sequences will be acquired in contiguous slices. The procedure will be followed on sedation and off sedation for healthy volunteers (in random order) and at mean arterial pressure of 65 mmHg and 75 mmHg (in random order) in patients receiving vasopressor therapy.

CONTACTS AND LOCATIONS:
Overall Officials: François Lamontagne, Principal Investigator — Université de Sherbrooke
Locations (1):
- Université de Sherbrooke, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided